CLINICAL TRIAL: NCT03804567
Title: Oldpain2go®: an Exploratory (Pre-Feasibility) Study.
Acronym: Oldpain2go®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Alasdair MacSween, Principal Lecturer in Research Governance, Teesside University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 163/18
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Pain, Chronic
Keywords: Oldpain2go®; Feasibility
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oldpain2go® (Experimental): This is a concept of dealing with a client in a way that uses their conscious mind to alter their unconscious automated programs (chronic pain) that are troubling them.
  Interventions: Other: Oldpain2go®
- Routine low back pain management (Active Comparator): Normal accepted physiotherapy treatment for persistent low back pain.
  Interventions: Other: Routine low back pain management

INTERVENTIONS:
Other: Oldpain2go® — This is a concept of dealing with a client in a way that uses their conscious mind to alter their unconscious automated programs such as chronic pain that are troubling them.
  Arms: Oldpain2go®
Other: Routine low back pain management — Standard low back persistent physiotherapy management as recommended by national guidelines.
  Arms: Routine low back pain management

SUMMARY:
Research question: Is there any evidence to suggest that the oldpain2go® intervention merits scientific investigation?

DETAILED DESCRIPTION:
Aims:

1. To collect data to:

   1. give an indication of the potential effect size, of any effects, from the oldpain2go® intervention, in people with persistent low back pain.
   2. to explore the eligibility criteria, recruitment methods and materials proposed here, for potential use in a future Feasibility study, of the oldpain2go® intervention.
2. To compare demographic characteristics, medical history and outcome measure data of:

   1. people for whom Oldpain2go® is indicated (at the Oldpain2go® screening session), with those for whom it is not,
   2. people for whom the Oldpain2go® intervention works, after one treatment, with those for whom it does not, and
   3. people for whom the Oldpain2go® intervention works, after one, or two, treatments, with those for whom it does not work after two treatments.

ELIGIBILITY:
Inclusion Criteria:

* Currently suffering from persistent, non-specific, low back pain
* Aged over 18 years
* For whom Oldpain2go® is indicated as a treatment option after the standard clinical screening process for the Oldpain2go® treatment

Exclusion Criteria:

* Any Red Flags,
* Any causative (or potentially causative) structural abnormality, or pathology detected or suspected
* Any concurrent pathology, or condition that would limit options for Physiotherapy treatment,
* Lack of (or any reason to doubt presence of) Mental Capacity to give Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
A 100mm pain intensity Visual Analogue Scale (VAS) for low back pain | Change measures at three points, baseline, 1 week and 2 weeks from baseline
  A self reported pain level scale

SECONDARY OUTCOMES:
The Roland Morris Disability Questionnaire (RMDQ) | Change measures at three points, baseline, 1 week and 2 weeks from baseline
  A measure of disability

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair MacSween, Dr, Principal Investigator — Teesside University
Locations (1):
- Norton Physiotherapy Centre, Norton, Stockton-on-Tees, United Kingdom